CLINICAL TRIAL: NCT05023720
Title: Real-World Effectiveness of Regorafenib in the Treatment of Patients With Metastatic Colorectal Cancer-A Retrospective Study
Brief Title: Real-World Effectiveness of Regorafenib in the Treatment of Patients With Metastatic Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Shujun Yang, Director, Henan Cancer Hospital
Other Study IDs: YShujun
Record Dates: First submitted 2021-07-29; First posted 2021-08-26 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Metastatic Colorectal Cancer
Keywords: metastatic colorectal cancer; regorafenib
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Regorafenib group: Patients were given only regorafenib orally
  Interventions: Other: nonintervention
- Joint group: The patient was treated with regorafenib orally and in combination with other medications
  Interventions: Other: nonintervention

INTERVENTIONS:
Other: nonintervention

SUMMARY:
Real-World Effectiveness of Regorafenib in the Treatment of Patients with Metastatic Colorectal Cancer- A Retrospective, Observational Study

DETAILED DESCRIPTION:
To analyze the real-world usage pattern, effectiveness and factors associated with the effectiveness of regorafenib in the treatment of patients with metastatic colorectal cancer (mCRC). This retrospective, observational study included clinicopathological and follow-up data of patients with mCRC who were treated with regorafenib from June 2017 to September 2020. Patients with incomplete data were excluded. Overall survival (OS) stratified by combination therapy with programmed cell death ligand-1 (PD-L1) inhibitors, chemotherapy and regorafenib dose was calculated by Kaplan Meier method and log rank test. R software version 4.0 was used for the analysis.

ELIGIBILITY:
1. Inclusion Criteria:

   1. Must be a pathologically proven colorectal adenocarcinoma
   2. Must have been treated with regorafenib
   3. Regorafenib must be used after two lines of standard antitumor therapy
2. Exclusion Criteria:

   1. Application is less than one course of treatment with regorafenib
   2. First - or second-line treatment with regorafenib
   3. Patients with multiple primary cancers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pathologically proven colorectal adenocarcinoma whose disease progressed after two lines of antitumor therapy were treated with regorafenib alone or in combination.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-07-20 (Actual); Primary Completion 2022-12-21 (Estimated); Study Completion 2022-12-21 (Estimated)

PRIMARY OUTCOMES:
The difference in overall survival between the two groups calculated by Kaplan-Meier | 2021.7-2022.12
  Survival differences between the monotherapy and combination groups
The difference of OS in patients receiving different doses of regorafenib | 2021.11-2022.12
  In the real world, regorafenib was used in different dosages: 40mg,80mg,120mg,160mg,respectively. The difference in overall survival time of patients with different dosage was compared.
Regorafenib in combination with other drugs | 2021.7-2022.10
  In the real world, regorafenib was used in combination with chemotherapy, immunotherapy or other drugs, and the frequency of occurrence of different conditions was analyzed.

SECONDARY OUTCOMES:
Survival differences among the patients with different clinical phenotypes and genotypes | 2021.7-2022.10
  To compare the survival of patients with mCRC by gender, age, tumor site and other genotypes

CONTACTS AND LOCATIONS:
Overall Officials: Shujun Yang, Study Director — Henan Cancer Hospital
Locations (1):
- Henan cancer hosiptal, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Yes
Clinical data of the patients
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: At any time
Access Criteria: Research needs